CLINICAL TRIAL: NCT00958698
Title: NURSE-DELIVERED WRITE SYMPTOMS vs. SELF-DIRECTED WRITE SYMPTOMS vs. CARE AS USUAL FOR OPTIMAL SYMPTOM MANAGEMENT FOR WOMEN WITH RECURRENT OVARIAN, FALLOPIAN TUBE, OR PRIMARY PERITONEAL CANCER
Brief Title: Symptom Management in Patients With Recurrent or Persistent Ovarian Cancer, Fallopian Tube Cancer, or Primary Peritoneal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GOG-0259; NCI-2011-01950 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000648729; GOG-0259 (Other: Gynecologic Oncology Group); GOG-0259 (Other: DCP); GOG-0259 (Other: CTEP); U10CA101165 (NIH)
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Fallopian Tube Carcinoma; Primary Peritoneal Carcinoma; Psychological Impact of Cancer; Recurrent Ovarian Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods; Psychiatric Rehabilitation

ARMS (3):
- Arm I (nurse-assisted intervention module) (Experimental): Patients are given password-protected access to their own web-based message board to communicate with a research nurse. The nurse leads patients through WRITE Symptoms? intervention module, with personalized support and advice. The nurse will encourage the patient to try new selected strategies, continue with effective strategies, and work with local health care providers in an ongoing process to improve symptom management.
  Interventions: Other: Communication Intervention; Other: Educational Intervention; Other: Internet-Based Intervention; Procedure: Psychosocial Assessment and Care; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (self-directed intervention module) (Experimental): Patients are given password-protected access to an interactive web-based computer program that will lead them through a modified WRITE Symptoms? intervention module (comprising the same elements as in arm I) without guidance and individualized recommendations from a nurse. Patients work through 3 selected symptoms using the WRITE Symptoms? intervention module over approximately 4 weeks. The program will generate an encouragement for the patient to try new selected strategies, continue with effective strategies, and continue the new approach to symptom management with local health care providers in an ongoing process to improve symptom management.
  Interventions: Other: Educational Intervention; Other: Internet-Based Intervention; Procedure: Psychosocial Assessment and Care; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm III (standard care from local provider) (Active Comparator): Patients are given password-protected access to online questionnaires. Patients are prompted monthly to complete online questionnaires. Patients receive standard symptom management from their local health care providers.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Communication Intervention — Ancillary studies
  Arms: Arm I (nurse-assisted intervention module)
Other: Educational Intervention — Ancillary studies
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Arm I (nurse-assisted intervention module); Arm II (self-directed intervention module)
Other: Internet-Based Intervention — Ancillary studies
  Arms: Arm I (nurse-assisted intervention module); Arm II (self-directed intervention module)
Procedure: Psychosocial Assessment and Care — Ancillary studies
  Other Names: Psychosocial Care/Assessment
  Arms: Arm I (nurse-assisted intervention module); Arm II (self-directed intervention module)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized clinical trial is studying two different symptom management programs to see how well they work compared with usual care in patients with recurrent or persistent ovarian cancer, fallopian tube cancer, or primary peritoneal cancer. Developing a symptom management plan may help relieve symptoms related to cancer or cancer treatment and help improve quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Compare the efficacy of nurse-delivered WRITE Symptoms? and self-directed WRITE Symptoms? vs usual care interventions in improving target symptom representations (i.e., decreases in symptom severity, symptom-related distress, and symptom consequences as measured by the Symptom Representation Questionnaire [SRQ]) in patients with recurrent or persistent ovarian, fallopian tube, or primary peritoneal cancer.

SECONDARY OBJECTIVES:

I. Compare the efficacy of nurse-delivered WRITE Symptoms? vs self-directed WRITE Symptoms? vs usual care interventions in improving target symptom representations in these patients at 4 weeks.

II. Compare the efficacy of nurse-delivered WRITE Symptoms? vs self-directed WRITE Symptoms? vs usual care interventions in improving target symptom controllability in these patients at 4, 8, and 12 weeks.

III. Compare the efficacy of nurse-delivered WRITE Symptoms? vs self-directed WRITE Symptoms? vs usual care interventions in improving indicators of quality of life (QOL) of these patients as measured by the FACT-O and the CES-Depression inventory short form at 4, 8, and 12 weeks.

IV. Compare the efficacy of nurse-delivered WRITE Symptoms? vs self-directed WRITE Symptoms? vs usual care interventions in improving communication with health care providers about symptoms, implementation of new symptom management strategies (health care provider recommended as well as patient-initiated changes), and perceived effectiveness of strategies (health care provider recommended as well as patient-initiated changes) in these patients at 4, 8, and 12 weeks.

V. Compare the efficacy of nurse-delivered WRITE Symptoms? vs self-directed WRITE Symptoms? vs usual care interventions in improving patient-related barriers to symptom management as measured by the Symptom Management Barriers Questionnaire at 4, 8, and 12 weeks.

EXPLORATORY OBJECTIVES:

I. Compare trajectories of change for overall symptom severity in patients undergoing nurse-delivered WRITE Symptoms? vs self-directed WRITE Symptoms? vs usual care interventions using monthly assessments to explore potential long-term effects of the WRITE Symptoms? interventions.

II. Compare trajectories of change for QOL of patients undergoing nurse-delivered WRITE Symptoms? vs self-directed WRITE Symptoms? vs usual care interventions using monthly assessments to explore potential long-term effects of the WRITE Symptoms? interventions.

III. Compare trajectories of change for symptom severity, distress, communication, and implementation of new strategies for non-targeted symptoms in patients undergoing nurse-delivered WRITE Symptoms? vs self-directed WRITE Symptoms? vs usual care interventions using monthly assessments to explore whether patients are able to generalize the symptom management approaches taught in WRITE Symptoms? interventions to their other non-targeted symptoms.

IV. Explore whether changes in symptom representations mediate changes in QOL of these patients at 8 and 12 weeks.

V. Explore whether effects of the WRITE Symptoms? interventions on primary and secondary endpoints at 8 and 12 weeks differ based on the following patient characteristics assessed at baseline: age, education, and ethnicity; depression as measured by the CES-D short form; trait anxiety as measured by the STAI; optimism as measured by the LOT-R; social support as measured by the ISEL; and symptom severity as measured by the SRQ.

OUTLINE: This is a multicenter study. Patients are stratified according to race/ethnicity (non-Hispanic white vs Hispanic or non-white). Patients are randomized to 1 of 3 intervention arms.

ARM I (nurse-delivered intervention): Patients are given password-protected access to their own web-based message board to communicate with a research nurse. The nurse leads the patient through the WRITE Symptoms? intervention module comprising representational assessment; exploring concerns/misconceptions/gaps/confusions; creating conditions for conceptual change; introducing new information, goal setting, and development of a symptom management plan; and summary via asynchronous postings to the patient's message board. Patients work through 3 selected symptoms using the nurse-delivered WRITE Symptoms? intervention module over approximately 4 weeks. Two weeks later, the patient's symptom management strategy and their desire to make further changes are evaluated by additional interaction with the nurse via the message board. The nurse will encourage the patient to try new selected strategies, continue with effective strategies, and work with local health care providers in an ongoing process to improve symptom management. Patients are given access to a resource guide that includes self-care guides for 26 symptoms. They are encouraged to use the same process taught for their 3 selected symptoms for any other symptoms that arise after the course of the intervention.

ARM II (self-directed intervention): Patients are given password-protected access to an interactive web-based computer program that will lead them through a modified WRITE Symptoms? intervention module (comprising the same elements as in arm I) without guidance and individualized recommendations from a nurse. Patients work through 3 selected symptoms using the WRITE Symptoms? intervention module over approximately 4 weeks. Two weeks later, patients are prompted by the computer program to respond to questions about their symptom management strategy and their desire to make further changes. The program will generate an encouragement for the patient to try new selected strategies, continue with effective strategies, and continue the new approach to symptom management with local health care providers in an ongoing process to improve symptom management. Patients are given access to a resource guide that includes self-care guides for 26 symptoms. They are encouraged to use the same process taught for their 3 selected symptoms for any other symptoms that arise after the course of the intervention.

ARM III (usual care): Patients are given password-protected access to online questionnaires. Patients are prompted monthly to complete online questionnaires. Patients receive standard symptom management from their local health care providers.

In all arms, patients complete online questionnaires to assess outcome measures at baseline, at 4, 8, and 12 weeks, and then every 4 weeks for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ovarian, fallopian tube, or primary peritoneal cancer that has recurred or persisted following primary therapy

  * Active disease or current treatment are not required
* Must be experiencing ? 3 symptoms associated with ovarian cancer or cancer treatment, including, but not limited to, any of the following:

  * Abdominal bloating or cramping
  * Nausea, vomiting, or diarrhea
  * Constipation
  * Anorexia
  * Anxiety
  * Depression
  * Dizziness
  * Drowsiness
  * Dry mouth
  * Fatigue
  * Headaches
  * Hair loss
  * Hot flashes
  * Memory concerns
  * Mood swings
  * Mouth sores
  * Pain
  * Peripheral neuropathies
  * Sexuality concerns
  * Sleep disturbances
  * Shortness of breath
  * Skin rash or palmar-plantar erythrodysesthesia
  * Urinary problems
  * Weight gain or loss
* GOG performance status 0-2
* Able to read and write English
* Access to computer and the Internet required
* Concurrent treatment on other clinical trials allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 485 (Actual)
Dates: Start 2010-01-19 (Actual); Primary Completion 2017-01-08 (Actual)

PRIMARY OUTCOMES:
Symptom severity, symptom-related distress, consequences, and control of symptoms as measured by the Symptom Representation Questionnaire | Baseline and at 4, 8, and 12 weeks

SECONDARY OUTCOMES:
Health-related quality of life as measured by the FACT-O | Baseline and at 4, 8, and 12 weeks, and every 4 weeks for 1 year
Depressive symptoms as measured by the CES-D short form | Baseline and at 4, 8, and 12 weeks, and every 4 weeks for 1 year
Communication with health care providers and use of self-care strategies assessed by investigator-developed survey | Baseline and at 4, 8, and 12 weeks
Implementation and perceived effectiveness of new symptom management strategies assessed by questionnaire | Baseline and at 4, 8, and 12 weeks
Barriers to symptom management as measured by the Symptom Management Barriers Questionnaire | Baseline and at 4, 8, and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Donovan, Principal Investigator — Gynecologic Oncology Group
Locations (144):
- United States (144):
  - Gynecologic Oncology Group of Arizona, Phoenix, Arizona
  - Cedars Sinai Medical Center, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - University of Colorado Hospital, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Queen's Medical Center, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Decatur Memorial Hospital, Decatur, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Providence Medical Center, Kansas City, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Shawnee Mission Medical Center-KCCC, Shawnee Mission, Kansas
  - CHRISTUS Highland Medical Center, Shreveport, Louisiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Massachusetts Memorial Health Care, Worcester, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - Memorial Medical Center - Las Cruces, Las Cruces, New Mexico
  - Island Gynecologic Oncology, Brightwaters, New York
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Main Line Health NCORP, Wynnewood, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - The Methodist Hospital System, Houston, Texas
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin

REFERENCES:
- [Derived] Donovan HS, Sereika SM, Wenzel LB, Edwards RP, Knapp JE, Hughes SH, Roberge MC, Thomas TH, Klein SJ, Spring MB, Nolte S, Landrum LM, Casey AC, Mutch DG, DeBernardo RL, Muller CY, Sullivan SA, Ward SE. Effects of the WRITE Symptoms Interventions on Symptoms and Quality of Life Among Patients With Recurrent Ovarian Cancers: An NRG Oncology/GOG Study (GOG-0259). J Clin Oncol. 2022 May 1;40(13):1464-1473. doi: 10.1200/JCO.21.00656. Epub 2022 Feb 7. PMID 35130043